CLINICAL TRIAL: NCT04230993
Title: Clinical Evaluation of the Efficacy of Two Nasal Products for Decongestion and Mucus Fluidification
Brief Title: Efficacy of Two Nasal Products for Decongestion and Mucus Fluidification
Acronym: DEFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YSLab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01705-52
Record Dates: First submitted 2020-01-03; First posted 2020-01-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ocean Bio Actif-Fluid+ (Experimental): Moderate hypertonic seawater solution (15 g / L NaCl) with polysorbate 80. The use is 1 to 2 sprays per nostril 4 times a day until symptoms of cold disappear, according to the instructions for use of the products.
  Interventions: Other: Sea water solution
- Ocean Bio Active-Stuffy nose (Experimental): Moderate hypertonic seawater solution (15 g / L NaCl) without polysorbate 80. The use is 1 to 2 sprays per nostril 4 times a day until symptoms of cold disappear, according to the instructions for use of the products.
  Interventions: Other: Sea water solution
- Ocean Bio Active-Hygiene of the nose (Active Comparator): Isotonic seawater solution (9 g / L NaCl). The use is 1 to 2 sprays per nostril 4 times a day until symptoms of cold disappear, according to the instructions for use of the products.
  Interventions: Other: Sea water solution

INTERVENTIONS:
Other: Sea water solution — Administration of different sea water solution is performed and the rating of cold symptoms according to the Jackson scale, the fluidity of mucus and the ease of blowing will be evaluated.

SUMMARY:
The main objective is to compare the effect of nasal washing on nasal discharge and nasal congestion during treatment after 3 days of use.

DETAILED DESCRIPTION:
The main endpoint is a symptom score derived from the Jackson scale: sum of 2 items relating to runny nose and nasal congestion (stuffy nose), with ratings of 0 to 3 for each (0: absent ; 1: mild; 2: moderate; 3: severe).

ELIGIBILITY:
Inclusion Criteria:

* Person with an upper respiratory condition (cold, rhinitis, nasopharyngitis ...) with symptoms of nasal congestion and intense runny nose moderate to severe (Jackson derived score ≥ 4)
* Ability of the patient (for adults) or their legal representative (for children) to follow the guidelines of the medical device
* have given their written informed consent

Exclusion Criteria:

* Patient with no cold symptoms, including no nasal congestion (chronic dry rhinitis…)
* Patient under treatment with cortisone derivative, mucolytic, or medication containing pseudoephedrine or related product acting on nasal congestion or having used such a product in the 3 days before inclusion
* Patient who used a nasal wash product in the 3 days before inclusion
* Patient allergic to seafood, or to any of the components of the products under study
* Vulnerable patient whose inclusion is not justified by the research objectives: woman pregnant, parturient, psychiatric patient, or adult subject to legal protection
* Patient participating or having participated in any other clinical study in the 30 days before the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Effect of nasal washing with a hypertonic seawater solution Nose hygiene). | 3 days
  Effect of nasal washing with a hypertonic seawater solution (Ocean Bio Actif-Fluid + or Ocean Bio Actif-Stuffy nose) on runny nose and nasal congestion during treatment after 3 days of use, compared to an isotonic solution (Ocean Bio Actif- Nose hygiene). symptom score (runny nose and nasal congestion) derived from the Jackson scale with a score of 0 to 3 for each (0: absent; 1: mild; 2: moderate; 3: severe) between Day 0 and Day 3.

SECONDARY OUTCOMES:
Symptom score | 7 days
  The effect of nasal wash on the evolution of symptoms over time
Presence or absence of fluid mucus | 7 days
  The effect of nasal wash on the evolution of the mucus fluidification over time
Global Clinical Impression Scale | between day 3 and day 7
  Global Clinical Impression of the investigator on the evolution of symptoms
Global Patient Impression Scale | between day 3 and day 7
  Global Impression of the patient on the evolution of symptoms
Use of medical device | 7 days
  Number of daily sprays
Safety of medical device | 7 days
  Number of adverse events
Likert scale | 7 days
  Satisfaction of patient for the medical device
Number of concomitant treatment | 7 days
  concomitant administration of treatments related to rhinitis

CONTACTS AND LOCATIONS:
Overall Officials: Alain BOYE, MD, Principal Investigator — Coordinator of the study
Locations (1):
- Medical office, Oignies, France

IPD SHARING:
Plan to Share IPD: No